CLINICAL TRIAL: NCT04670900
Title: Operative or Non-Operative Treatment of Displaced Fractures of the Elderly - a Nordic Multicenter Randomized Trial
Brief Title: Treatment of Olecranon Fractures in the Elderly
Acronym: CROFT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Frede Frihagen, Associate professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC2018/88
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Olecranon Fracture
Keywords: Elderly patients; Surgery; Non-operative treatment; Functional outcome
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Intervention Model Description: Randomized non-inferiority multicenter
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patient instructed not to reveal treatment and to wear long sleeves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operative (Active Comparator): Patients will be operated according to Orthopedic Trauma Association (OTA) principles with either tension band wiring or plate fixation with an anatomical precontoured plate.
  Interventions: Procedure: Tension band wiring or plate fixation
- Non-operative (Experimental): Patients will be offered a plaster cast for 1-2 weeks
  Interventions: Procedure: Active non-operative treatment with optional plaster cast

INTERVENTIONS:
Procedure: Tension band wiring or plate fixation — Choice of operative treatment is TBW or PF with a precontoured anatomical plate. The treating surgeon decides if TBW or PF is chosen as operative treatment method. The surgeries are performed according to OTA principles by an experienced surgeon, a trauma fellow or a consultant as approved by the participating hospitals.
  Arms: Operative
Procedure: Active non-operative treatment with optional plaster cast — Patients allocated to non-operative treatment are offered a back-slab in 60 degrees of flexion for pain-relief. The back-slab is removed 7-14 days following injury.
  Arms: Non-operative

SUMMARY:
Operative treatment, with tension band wiring or plate fixation, will be compared with non-operative treatment of displaced olecranon fractures (Mayo classification 2A and 2B) in patients 75 years or older.

DETAILED DESCRIPTION:
Displaced olecranon fractures disrupt the extensor mechanism of the elbow and operative treatment is therefore usually recommended. Tension band wiring (TBW) and plate fixation (PF) are the most common surgical treatment options. Both methods are associated with high complication and reoperation rates, especially in elderly patients. Only one randomized controlled trial has compared operative and non-operative treatment of olecranon fractures in the elderly, but the study was stopped prematurely due to high complication rates in the group treated operatively and remained underpowered for important outcome measures.A few small patient series with non-operatively treated fractures also exist and suggest that it may be a valid alternative to operative treatment

ELIGIBILITY:
Inclusion Criteria:

* Displaced olecranon fracture (Mayo 2A and 2B).

Exclusion Criteria:

* Associated fractures in the coronoid process, radial head or distal humerus.
* Open fracture, Gustilo-Andersen 2 or 3
* Severe cardiopulmonary disease or other medical condition which contraindicates surgery.
* Previous injury to or other condition in the elbow with serious functional impairment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Oxford Elbow Score | 52 weeks
  Patient reported 12 item form, 0 (worst) to 100 (best possible score)

SECONDARY OUTCOMES:
Range of motion | 6 weeks
  Extension, flexion, rotation
Range of motion | 12 weeks
  Extension, flexion, rotation
Range of motion | 52 weeks
  Extension, flexion, rotation measured in degrees total movement for each direction.
Elbow extension strength | 6 weeks
  Strength measured isometrically on a scale (grams) with elbow in 30 degrees flexion. Both arms measured for comparison.
Elbow extension strength | 12 weeks
  Strength measured isometrically on a scale (grams) with elbow 30 degrees flexion. Both arms measured for comparison.
Elbow extension strength | 52 weeks
  Strength measured isometrically on a scale (grams) with elbow 30 degrees flexion. Both arms measured for comparison. arms measured for comparison.
Elbow satisfaction | 6 weeks
  Single question: Are you satisfied with your elbow? Yes/Somewhat/No
Elbow satisfaction | 12 weeks
  Single question: Are you satisfied with your elbow? Yes/Somewhat/No
Elbow satisfaction | 52 weeks
  Single question: Are you satisfied with your elbow? Yes/Somewhat/No
Complications | Through study period up to 52 weeks.
  Serious local complications not reoperated.
Number of Reoperations | Through study period up to 52 weeks.
  Any reoperation
Oxford Elbow Score | 6 weeks
  Patient reported 12 item form, 0 (worst) to 100 (best possible score)
Oxford Elbow Score | 12 weeks
  Patient reported 12 item form, 0 (worst) to 100 (best possible score)

CONTACTS AND LOCATIONS:
Overall Officials: Frede Frihagen, PhD, Principal Investigator — University of Oslo
Locations (12):
- Norway (11):
  - Baerum Hospital, Sandvika, Gjettum
  - Vestre Viken Hospital Trust, Hønefoss, Norway
  - St. Olavs Hospital, Trondheim, Trønderlag
  - Arendal Hospital, Arendal
  - Haukeland University Hospital, Bergen
  - Østfold Hospital Trust, Grålum
  - Orthopedic Center, Ulleval University Hospital, Oslo
  - Diakonhjemmet Hospital, Oslo
  - Telemark Hospital, Skien
  - Stavanger University Hospital, Stavanger
  - Tønsberg Hospital, Tønsberg
- Akademiska Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Publish protocol
Supporting Information: Study Protocol
Time Frame: Within 12 months
Access Criteria: Open access

REFERENCES:
- [Background] Savvidou OD, Koutsouradis P, Kaspiris A, Naar L, Chloros GD, Papagelopoulos PJ. Displaced olecranon fractures in the elderly: outcomes after non-operative treatment - a narrative review. EFORT Open Rev. 2020 Aug 1;5(7):391-397. doi: 10.1302/2058-5241.5.190041. eCollection 2020 Jul. PMID 32818066